CLINICAL TRIAL: NCT04175665
Title: Semaglutide in Patients With Type 2 Diabetes: Real-world Analysis in the Canadian LMC Diabetes Registry: The SPARE Study
Brief Title: Real-world Health Outcomes in Canadian Patients Using Semaglutide
Status: Completed | Type: Observational
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: SPARE
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes
Keywords: semaglutide; retrospective study; hemoglobin A1c; body weight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Body Weight | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Semaglutide — Prescription for semaglutide as part of usual clinical practice
  Other Names: Ozempic

SUMMARY:
Glucagon-like peptide-1 receptor agonists (GLP-1 RA) are an injectable, non-insulin therapy for patients with type 2 diabetes (T2D). Semaglutide (Ozempic®) is the newest GLP-1 RA to become available in Canada in 2018, and is administered subcutaneously once-weekly. In clinical trials, semaglutide has been superior to placebo and other antihyperglycemic agents in HbA1c reduction and body weight loss. However, there is little real-world evidence available on the effectiveness of semaglutide in real-world clinical practice.

To better understand the effectiveness of semaglutide on clinical outcomes in a real-world setting, this retrospective cohort study will use the Canadian LMC Diabetes Registry to examine the effects of semaglutide on glycemic control, body weight, and other clinical outcomes in patients with T2D who initiate once-weekly semaglutide as part of usual clinical care in a diabetes specialist practice group in Canada.

ELIGIBILITY:
Inclusion Criteria:

* First prescription for semaglutide between Feb 1 2018 and Feb 1 2019
* Age ≥ 18 years at medication index date
* Clinical diagnosis of type 2 diabetes for greater than six months
* ≥ one HbA1c measurement at baseline and at follow-up
* ≥ one follow-up visit post index date
* Informed consent for medical data to be used for research purposes

Exclusion Criteria:

* Clinical diagnosis of type 1 diabetes
* Recent eGFR <40 ml/min/1.73m2
* Documented history of bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients with type 2 diabetes who initiate semaglutide between February 1, 2018 and February 1, 2019 as part of usual clinical care, and who are active patients at LMC Diabetes & Endocrinology.
Sampling Method: Non-Probability Sample
Enrollment: 1133 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-02-09 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 3 to 6 months
  Change in HbA1c (%) between baseline and last measured value at 3 to 6 months follow-up

SECONDARY OUTCOMES:
Change in body weight | 3 to 6 months
  Change in body weight (kg) between baseline and last measured value at 3 to 6 months follow-up
Change in body mass index (BMI) | 3 to 6 months
  Change in BMI (kg/m2) between baseline and last measured value at 3 to 6 months follow-up
Change in systolic blood pressure (SBP) | 3 to 6 months
  Change in SBP (mmHg) between baseline and last measured value at 3 to 6 months follow-up
Change in diastolic blood pressure (DBP) | 3 to 6 months
  Change in DBP (mmHg) between baseline and last measured value at 3 to 6 months follow-up
Change in triglycerides | 3 to 6 months
  Change in triglycerides (mmol/L) between baseline and last measured value at 3 to 6 months follow-up
Change in LDL cholesterol | 3 to 6 months
  Change in LDL cholesterol (mmol/L) between baseline and last measured value at 3 to 6 months follow-up
Change in non-HDL cholesterol | 3 to 6 months
  Change in non-HDL cholesterol (mmol/L) between baseline and last measured value at 3 to 6 months follow-up
Change in estimated glomerular filtration rate (eGFR) | 3 to 6 months
  Change in eGFR (mL/min/1.73 m2) between baseline and last measured value at 3 to 6 months follow-up
Change in alanine amino transaminase (ALT) | 3 to 6 months
  Change in ALT (U/L) between baseline and last measured value at 3 to 6 months follow-up
Proportion of patients who report ≥ 1 weekly incidence of any hypoglycemia | 3 to 6 months
  Analyses will also be stratified by sulfonylurea (SU) versus non-SU use, and insulin versus non-insulin use
Proportion of patients who report ≥ 1 yearly incidence of severe hypoglycemia | 3 to 6 months
  Analyses will also be stratified by SU versus non-SU use, and insulin versus non-insulin use
Proportion of patients who achieve HbA1c ≤7.0% | 3 to 6 months
  HbA1c will be the last measured value at 3 to 6 months follow-up
Proportion of patients who achieve HbA1c ≤8.0% | 3 to 6 months
  HbA1c will be the last measured value at 3 to 6 months follow-up
Proportion of patients who achieve HbA1c reduction ≥0.5% | 3 to 6 months
  HbA1c will be the last measured value at 3 to 6 months follow-up
Proportion of patients who achieve HbA1c reduction ≥1.0% | 3 to 6 months
  HbA1c will be the last measured value at 3 to 6 months follow-up
Proportion of patients who achieve weight loss ≥5% | 3 to 6 months
  Weight will be the last measured value at 3 to 6 months follow-up
Proportion of patients who achieve weight loss ≥10% | 3 to 6 months
  Weight will be the last measured value at 3 to 6 months follow-up

OTHER OUTCOMES:
Time to addition of another diabetes therapy | 3 to 6 months
  Number of weeks until addition of another diabetes therapy
Time to discontinuation of GLP-1 RA therapy | 3 to 6 months
  Number of weeks until discontinuation of semaglutide therapy in patients who discontinue semaglutide during the follow-up period
Insulin dose at baseline and follow-up | 3 to 6 months
  Insulin dose will be evaluated in the subgroup of patients using insulin therapy
HbA1c change in low dose therapy and high dose therapy subgroups | 3 to 6 months
  Low dose therapy (semaglutide 0.5 mg) and full dose therapy (semaglutide 1.0 mg)
Body weight change in low dose therapy and high dose therapy subgroups | 3 to 6 months
  Low dose therapy (semaglutide 0.5 mg) and full dose therapy (semaglutide 1.0 mg)
HbA1c change in patients who discontinue a dipeptidyl peptidase-4 inhibitor (DPP-4i) at baseline versus simple addition of semaglutide | 3 to 6 months
Body weight change in patients who discontinue a DPP-4i at baseline versus simple addition of semaglutide | 3 to 6 months
HbA1c change in patients who discontinue any diabetes therapy at baseline versus simple addition of semaglutide | 3 to 6 months
Body weight change in patients who discontinue any diabetes therapy at baseline versus simple addition of semaglutide | 3 to 6 months
HbA1c change in insulin users and non-insulin users | 3 to 6 months
  Based on insulin therapy used at baseline
Weight change in insulin users and non-insulin users | 3 to 6 months
  Based on insulin therapy used at baseline
HbA1c change in patients who have a 13-week follow-up versus a 26-week follow-up | 3 to 6 months
Weight change in patients who have a 13-week follow-up versus a 26-week follow-up | 3 to 6 months
HbA1c change in patients prescribed semaglutide as second line therapy (excluding insulin use) | 3 to 6 months
  In the subgroup of patients using one oral diabetes therapy at baseline
Weight change in patients prescribed semaglutide as second line therapy (excluding insulin use) | 3 to 6 months
  In the subgroup of patients using one other diabetes therapy at baseline
HbA1c change in patients prescribed semaglutide as third line therapy (excluding insulin use) | 3 to 6 months
  In the subgroup of patients using two oral diabetes therapies at baseline
Weight change in patients prescribed semaglutide as third line therapy (excluding insulin use) | 3 to 6 months
  In the subgroup of patients using two oral diabetes therapies at baseline
HbA1c change in patients prescribed semaglutide as fourth line therapy (excluding insulin use) | 3 to 6 months
  In the subgroup of patients using three oral diabetes therapies at baseline
Weight change in patients prescribed semaglutide as fourth line therapy (excluding insulin use) | 3 to 6 months
  In the subgroup of patients using three oral diabetes therapies at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Aronson, MD, Principal Investigator — LMC Diabetes & Endocrinology
Locations (1):
- LMC Diabetes & Endocrinology, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No